CLINICAL TRIAL: NCT01583179
Title: Duration of Analgesic Effect for Ultrasound Guided Supraclavicular Blocks With the Addition of Buprenorphine to Local Anesthetic Solution
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed prematurely due to low enrollment and anticipation of future barriers in enrollment
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-0781; SMPH/ANESTHESIO (Other: UW, Madison); A530900 (Other: UW, Madison)
Record Dates: First submitted 2012-04-19; First posted 2012-04-23 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Regional Block for Pain Control; Supraclavicular Block; Ultrasound Guided Block; Block Additive
Keywords: nerve block; outpatient surgery
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): will get only local anesthetic and epinephrine in block. no additive in block
- buprenorphine (Experimental): will receive local anesthetic, epinephrine and the additive buprenorphine to nerve block
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — added to nerve block, 0.3mg one time peripheral block use
  Arms: buprenorphine

SUMMARY:
The patients included will be those who have already agreed to have a brachial plexus nerve block for surgery. A flip of the coin will decide who gets and additive called buprenorphine in their block or not. They will both contain the same amount and type of numbing medicine. The goal will be to see if the additive extends the life of the pain control portion of the ultrasound guided supraclavicular nerve block.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1-3
2. Age 18-79, inclusive
3. BMI <36 kg/m^2
4. Patient consenting to single injection brachial plexus nerve block as primary anesthetic for a procedure

Exclusion Criteria:

1. Patients with coagulation disorders
2. Clinically significant pulmonary disease
3. Clinically significant cardiac disease
4. Neurologic deficit in surgical extremity
5. Allergy to bupivacaine or buprenorphine
6. Intolerance of narcotics
7. Local infection over intended area of needle insertion
8. Hepatic failure or renal failure
9. Significant psychiatric disease, including drug abuse
10. Seizure disorder
11. Possible pregnancy or lactation by patient report
12. Use of narcotic medication greater than 2 times a week for greater than 1 week.
13. Patients for whom the surgeon requests a shorter-acting block

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Donnelly, MD, Principal Investigator — University of Wisconsin School of Medicine and Public Health, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Buprenorphine
Started | 14 | 12
Completed | 13 | 10
Not Completed | 1 | 2
Not completed — Screen failure | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Buprenorphine | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Customized [Count of Participants; unit: Participants]
  Age of participants: 20-29 | 3 | 3 | 6
  Age of participants: 30-39 | 0 | 2 | 2
  Age of participants: 40-49 | 4 | 1 | 5
  Age of participants: 50-59 | 3 | 3 | 6
  Age of participants: 60-69 | 3 | 2 | 5
  Age of participants: 70-79 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 11 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time Until First Pain Medication Post-operatively
Description: Time in minutes until first pain medication was take by participant post-operatively
Time Frame: 48 hrs
Population: The study was closed prematurely due to low enrollment and anticipation of future barriers in enrollment.The Overall Number of Participants Analyzed represents the Number of Participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Time in minutes
Arm/Group | Control Group | Buprenorphine
Number analyzed (Participants) | 9 | 10
Time in minutes | 965 (250) | 862 (311)

2. Secondary Outcome: Pain Score on Post Operative Day 1
Description: pain score on post operative day 1 was measured on a scale 1-10. higher scores correlates with more severe pain. score range is from '0' (no pain) to 10 (pain as severe as it can be)
Time Frame: 1 day postoperative
Population: The study was closed prematurely due to low enrollment and anticipation of future barriers in enrollment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Buprenorphine
Number analyzed (Participants) | 10 | 12
score on a scale | 6.5 [4.25 to 7.75] | 4.5 [1.75 to 8.25]

ADVERSE EVENTS:
Description: Adverse events were not monitored. The study was closed prematurely due to low enrollment and anticipation of future barriers in enrollment
Arm/Group | Control Group | Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No